CLINICAL TRIAL: NCT07037459
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Maridebart Cafraglutide on Mortality and Morbidity in Participants Living With Heart Failure With Preserved or Mildly Reduced Ejection Fraction and Obesity (MARITIME-HF)
Brief Title: Maridebart Cafraglutide in Heart Failure With Preserved or Mildly Reduced Ejection Fraction and Obesity
Acronym: MARITIME-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230227
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Failure With Mildly Reduced Ejection Fraction; Obesity
Keywords: Heart Failure; Obesity; Maridebart Cafraglutide; AMG 133; MariTide
MeSH Terms: conditions — Obesity; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide (Experimental): Participants will receive maridebart cafraglutide subcutaneously (SC)
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
This trial will examine if maridebart cafraglutide as an adjunct to standard of care will lead to a reduction in heart failure (HF) events such as HF hospitalizations and urgent HF visits, cardiovascular (CV) deaths and improvement in HF symptoms in participants with HF with preserved ejection fraction (HFpEF) and HF with mildly reduced ejection fraction (HFmrEF) who are obese. This is a phase 3, global, multicenter, 2-part trial with a double-blind period and an open-label extension (OLE). The trial is event-driven, and Part 1 will conclude when approximately 850 primary endpoint events have occurred.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent.
* BMI ≥ 30.0 kg/m^2 at the time of randomization.
* HF diagnosed for at least 30 days with New York Heart Association (NYHA) Class II-IV at the time of informed consent.
* Managed with HF standard of care therapies.
* Left ventricular ejection fraction (LVEF) of > 40% within 12 months from the beginning of screening.
* Elevated NT-proBNP.
* Participants must have at least one of the following:

  1. Structural heart disease within 12 months prior to screening OR
  2. Documented hospitalization with a primary diagnosis of decompensated HF which required IV loop diuretic treatment > 30 days and < 12 months prior to randomization OR
  3. Evidence of elevated filling pressures within 12 months before randomization.

Exclusion Criteria:

* History of any of the following within 60 days prior to or during screening: Type I (spontaneous) MI, valvular replacement or repair, coronary revascularization, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke.
* HF due to: hypertrophic cardiomyopathy, infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac tamponade, arrhythmogenic right ventricular or left ventricular cardiomyopathy/dysplasia, uncorrected primary valvular heart disease, clinically significant congenital heart disease.
* Any lifetime history of LVEF ≤ 40%.
* Hospitalized with acute decompensated HF at the time of or during the screening period.
* Type 1 diabetes mellitus, or any type of diabetes with the exception of T2DM or history of gestational diabetes.
* For participants with a prior diagnosis of T2DM (including those diagnosed during screening):

  1. HbA1c > 10.0% (86 mmol/mol) at screening
  2. Uncontrolled diabetes requiring immediate therapy
  3. History of diabetic ketoacidosis or hyperosmolar state/coma within 12 months before randomization
  4. One or more episodes of severe hypoglycemia within 6 months before randomization and/or history of hypoglycemia unawareness
  5. History or presence of either proliferative diabetic retinopathy, or diabetic maculopathy, or severe non-proliferative diabetic retinopathy; or currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema.
* SBP ≥ 180 mmHg during the screening period, or on three or more blood pressure-lowering drugs with a SBP > 160 mmHg during the screening period.
* History of chronic pancreatitis or acute pancreatitis in the 180 days before screening or during the screening period.
* Any personal lifetime history of, or family history(first-degree relative[s]) of medullary thyroid carcinoma or MEN-2.
* eGFR < 20 mL/min/1.73 m^2 (CKD-EPI creatinine (Cr)-cystatin C equation) or receiving dialysis at screening.
* Calcitonin ≥ 50 ng/L (pg/mL) at screening.
* Acute or chronic hepatitis.
* Any of the following psychiatric history:

  1. History of unstable major depressive disorder or other severe psychiatric disorder within 2 years prior to screening or during the screening period
  2. Lifetime history of suicide attempt
  3. History of non-suicidal self-injury within 5 years prior to screening or during the screening period.
* History of any other condition that, in the opinion of the investigator, may preclude the participant from following the protocol and completing the trial.
* Use of any glucagon-like peptide 1 receptor agonist (GLP-1 RA), glucose-dependent insulinotropic polypeptide (GIP) agonists or antagonists, or amylin analogs within 90 days prior to or during the screening period or planned use during the conduct of the trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5056 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-09-29 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death or HF Events | Up to approximately 35 months
  Heart Failure events include: hospitalization for HF or urgent HF visits.

SECONDARY OUTCOMES:
Change From Baseline in Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score (CSS) for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Change from Baseline in the KCCQ Total Symptom Score (TSS) for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-TSS assesses symptom frequency and burden, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Total Number of HF Events Including First and Recurrent HF Events | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of: Myocardial Infarction (MI), Ischemic Stroke, CV Death (Major Adverse Cardiac Events [MACE]), or HF Events | Up to approximately 35 months
Time to First Event of a Composite Nephropathy Endpoint | Up to approximately 35 months
  The composite nephropathy endpoint consists of: persistent macroalbuminuria, persistent ≥ 40% reduction in estimated glomerular filtration rate (eGFR), onset of persistent eGFR < 15 mL/min/1.73 m^2, initiation of chronic renal replacement therapy (dialysis or transplantation), CV or renal death.
Change in eGFR Slope (Total) | Baseline up to approximately 35 months
Change in eGFR Slope (Chronic) | From 4 months up to approximately 35 months
Time to Onset of Type 2 Diabetes Mellitus (T2DM) in Participants with Prediabetes | Up to approximately 35 months
Time to the First HF Event | Up to approximately 35 months
Change from Baseline in the Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) | Baseline and Week 72
Change from Baseline in Body Mass Index (BMI) (kg/m^2) | Baseline and Week 72
Change from Baseline in the Waist Circumference (cm) | Baseline and Week 72
Change from Baseline in the Urine Albumin-to-creatinine Ratio (uACR) | Baseline and Week 72
Change from Baseline in the Hemoglobin A1c (HbA1c [%, mmol/mol]) in Participants with T2DM | Baseline and Week 72
Percent Change from Baseline in the High-sensitivity C Reactive Protein (hs-CRP) | Baseline and Week 72
Percent Change from Baseline in the Body Weight (kg) | Baseline and Week 72
Percent Change from Baseline in Total Cholesterol | Baseline and Week 72
Percent Change from Baseline in Non-high-density Lipoprotein Cholesterol (non-HDL-C) | Baseline and Week 72
Percent Change from Baseline in Low-density Lipoprotein Cholesterol (LDL-C), HDL-C, Triglycerides (TG), Very Low-density Lipoprotein Cholesterol (VLDL-C) | Baseline and Week 72
Total All-cause Hospitalizations (First and Recurrent Time to Event) | Up to approximately 35 months
Number of Participants Achieving ≥ 5-point Change in KCCQ-CSS Score from Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Number of Participants Achieving ≥ 10-point Change in KCCQ-CSS Score from Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Number of Participants Achieving an Anchor-based Change in KCCQ-CSS Score From Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life. The Patient Global Impression of Severity (PGI-S) and Patient Global Impression of Change (PGI-C) can be used as anchors to estimate within-patient change in the KCCQ-CSS score.
Number of Participants Achieving ≥ 5-point Change in KCCQ-TSS Score from Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-TSS assesses symptom frequency and burden, ranging from 0 to 100, with higher scores indicating better functioning and quality of life. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Number of Participants Achieving ≥ 10-point Change in KCCQ-TSS Score from Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-TSS assesses symptom frequency and burden, ranging from 0 to 100, with higher scores indicating better functioning and quality of life. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life.
Number of Participants Achieving an Anchor-based Change in KCCQ-TSS Score from Baseline for Participants with Baseline KCCQ-CSS Score ≤ 80 | Baseline and Week 48
  The KCCQ is a 23-item disease-specific measure for participants with HF, measuring the participant's perception of their health status. The KCCQ-TSS assesses symptom frequency and burden, ranging from 0 to 100, with higher scores indicating better functioning and quality of life. The KCCQ-CSS assesses symptoms and physical limitations, ranging from 0 to 100, with higher scores indicating better functioning and quality of life. The PGI-S and PGI-C can be used as anchors to estimate within-patient change in the KCCQ-CSS score.
Time to All-cause Death | Up to approximately 35 months
Time to CV Death | Up to Approximately 35 Months
Number of Participants with Treatment-emergent Adverse Events and Serious Adverse Events | Up to approximately 35 months
Plasma Concentration of Maridebart Cafraglutide | Week 72
Change from Baseline in N-terminal Pro B Type Natriuretic Peptide (NT-proBNP) | Baseline and Week 72
Time to New Onset of Atrial Fibrillation (AF) or Atrial Flutter (AFL) in Participants Without a History of AF or AFL at Baseline | Baseline and up to approximately 35 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (540):
- United States (96):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - SEC Clinical Research, Dothan, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - HonorHealth, Phoenix, Arizona
  - Medical Advancement Centers of Arizona, Phoenix, Arizona
  - Pima Heart and Vascular Clinical Research, Tucson, Arizona
  - Yuma Clinical Trials, Yuma, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - National Heart Institute, Beverly Hills, California
  - Valley Clinical Trials, LLC dba Flourish Research, Covina, California
  - National Institute of Clinical Research, Huntington Beach, California
  - 310 Clinical Research, Inglewood, California
  - Radin Cardiovascular Medical Group, Newport Beach, California
  - Valley Clinical Trials, Northridge, California
  - University of California Irvine, Orange, California
  - Empire Clinical Research, Pomona, California
  - San Diego Cardiac Center, San Diego, California
  - NorthBay Clinical Research LLC, Santa Rosa, California
  - Manshadi Heart Institute, Stockton, California
  - Cardiology Associates of Fairfield County PC, Stamford, Connecticut
  - Orlando Heart and Vascular Institute, Altamonte Springs, Florida
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Cardiovascular and Vein Center of Florida, Bradenton, Florida
  - Millennium Medical Research, Coral Gables, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - First Coast Cardiovascular Institute PA, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clearwater Cardiovascular Consultants, Largo, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Orlando Health Heart Institute, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Broward Research Center, Pembroke Pines, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Guardian Research Organization LLC, Winter Park, Florida
  - Privia Medical Group Georgia LLC, Peachtree City, Georgia
  - High Desert Heart and Vascular, Meridian, Idaho
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Midwest Cardiovascular Research And Education Foundation, Elkhart, Indiana
  - Ascension Medical Group, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Johnson County Clintrials, Lenexa, Kansas
  - Kansas Nephrology Research Institute LLC, Wichita, Kansas
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - Louisiana Heart Center - Hammond, Covington, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Northshore Heart and Vascular LLC, Mandeville, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants LLC, Beltsville, Maryland
  - Flourish Bowie, Bowie, Maryland
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Advanced Cardiology Associates, Rochester Hills, Michigan
  - Fairview Health Services M Health Fairview St Johns Hospital, Maplewood, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Bryan Heart, Lincoln, Nebraska
  - Methodist Physicians Clinic Heart Consultants, Omaha, Nebraska
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Virtua Health Incorporated, Marlton, New Jersey
  - CardioMetabolic Collaborative Clinic, Somerset, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Hudson Valley Cardiovascular Practice PC, Poughkeepsie, New York
  - Richmond University Medical Center, Staten Island, New York
  - Duke University Health System, Durham, North Carolina
  - Accellacare of Wilmington, Wilmington, North Carolina
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Abington Medical Specialists, Horsham, Pennsylvania
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Apex Research Foundation, LLC, Jackson, Tennessee
  - The Jackson Clinic PA, Jackson, Tennessee
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Cardiovascular Research of Knoxville North Knoxville Medical Center, Powell, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Javara Research, Conroe, Texas
  - Dallas Heart and Vascular Consultants, Duncanville, Texas
  - David Turbay, MD, El Paso, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Biopharma Informatic, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Vital Heart and Vein, Humble, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - Sherman Clinical Research, Sherman, Texas
  - Northwest Houston Clinical Research PLLC, Tomball, Texas
  - Carient Heart and Vascular, Manassas, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Pulse Heart Institute, Puyallup, Washington
- Argentina (20):
  - Imoba Investigaciones medicas, CABA, Buenos Aires
  - Centro de Investigaciones Metabolicas Cinme, CABA, Buenos Aires
  - Cemedic Centro de Especialidades Medicas, CABA, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, CABA, Buenos Aires
  - Fundacion Respirar - Consultorios Medicos Dr Doreski, CABA, Buenos Aires
  - Cardiología Palermo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Ciprec Centro de Investigacion y Prevencion Cardiovascular, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Mautalen Salud e Investigacion Expertia SA-Osteo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Ciad - Consultorio Integral de Atencion al Diabetico, Morón, Buenos Aires
  - Dim Clinica Privada, Ramos Meija, Buenos Aires
  - Go Centro Medico San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Clinica Fusavim Privada SRL, Villa María, Córdoba Province
  - Instituto de Investigaciones Clínicas Rosario-Sanatorio Delta, Rosario, Santa Fe Province
  - Instituto CAICI - Centro de Asistencia e Investigacion Clinica Integral, Rosario, Santa Fe Province
  - Centro Modelo de Cardiologia, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Instituto Medico Damic, Córdoba
  - INECO Neurociencias Oronio, Rosario
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
  - Instituto de Investigaciones Clinicas Zarate, Zárate
- Australia (15):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Sydney Cardiometabolic Centre, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Advara HeartCare Wesley, Auchenflower, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Gold Coast Hospital and Health Service, Southport, Queensland
  - Dr Heart Pty Ltd, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Victorian Heart Hospital, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Advara HeartCare Mulgrave, Mulgrave, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
- Austria (9):
  - Krankenhaus Sankt Josef Braunau, Braunau am Inn
  - Medizinische Universitaet Graz, Graz
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - Universitaetsklinikum Sankt Poelten, Sankt Pölten
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Ordinationszentrum imedneunzehn privat, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (15):
  - Azorg Campus Aalst - Moorselbaan, Aalst
  - Universitair Ziekenhuis Brussel, Brussels
  - Algemeen Ziekenhuis Sint Blasius, Dendermonde
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - AZ Herentals, Herentals
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Centre Hospitalier Chrétien MontLégia, Liège
  - AZ Delta Campus Rumbeke, Roeselare
  - Algemeen Ziekenhuis Turnhout, Turnhout
  - Universite Catholique de Louvain Cliniques Universitaires de Mont-Godinne, Yvoir
- Brazil (16):
  - Centro do Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Ccih - Consultoria em Controle de Infecção Hospitalar, Belo Horizonte, Minas Gerais
  - Cardresearch Cardiologia Assistencial de Pesquisa, Belo Horizonte, Minas Gerais
  - Nucleo de Pesquisa Clinica, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - jmf Clinica do Coracao ltda, Aracaju, Sergipe
  - Instituto de Pesquisa Clinica de Campinas - Ipecc, Campinas, São Paulo
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda - Clinica Loema, Campinas, São Paulo
  - Instituto do Coracao de Marilia, Marília, São Paulo
  - Clinicor Clinica Cardiologica, Ribeirão Preto, São Paulo
  - Pesquisare Saude Ltda, Santo André, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Bulgaria (13):
  - Ambulatory for special outpatient medical aid in Cardiology-Private Practice Dr Elena Dotcheva EOOD, Burgas
  - Multiprofile Hospital for Active Treatment - Haskovo AD, Haskovo
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Medical Center Futuremeds EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Knyaginya Klementina - Sofia EAD, Sofia
  - National Multiprofile Transport Hospital Tzar Boris III, Sofia
  - Multiprofile Hospital for Active Treatment National Hospital of Cardiology EAD, Sofia
  - Diagnostic-Consultative Center Alexandrovska EOOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Diagnostic-Consultative Center XX-Sofia EOOD, Sofia
  - Diagnostic-Consultative Center Convex OOD, Sofia
  - Multiprofile Regional Hospital for Active Treatment Dr Stefan Cherkezov AD, Veliko Tarnovo
  - Specialised Hospital for Active Cardiology Treatment EAD, Yambol
- Canada (19):
  - St Boniface Hospital, Winnipeg, Manitoba
  - Cardio 1, Winnipeg, Manitoba
  - Brampton Clinical Trials, Brampton, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Saul Vizel Professional Medicine Corporation - Vizel Cardiac Research, Cambridge, Ontario
  - Partners in Advanced Cardiac Evaluation, Newmarket, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - CardioQuest Research Centre, Sarnia, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - KMH Cardiology Centres Incorporated Hamilton, Stoney Creek, Ontario
  - Curans Heart Center, Thunder Bay, Ontario
  - Womens College Hospital, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Winchester District Memorial Hospital, Winchester, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Diex Recherche Sherbrooke Est, Sherbrooke, Quebec
  - Diex Recherche Trois Rivieres, Trois-Rivières, Quebec
- China (47):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Inner Mongolia Medical University, Haikou, Hainan
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Luoyang Third Peoples Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Peoples Hospital of Hubei Province, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - Hebei General Hospital, Hengyang, Hunan
  - First Affiliated Hospital of Baotou Hospital, Inner, Baotou, Inner Mongolia
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang Peoples Hospital, Pingxiang, Jiangxi
  - Jilin Province Peoples Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - China Japan Union Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Siping City Center Peoples Hospital, Siping, Jilin
  - Zhongshan Hospital Affiliated to Dalian University, Shenyang, Liaoning
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi An Medical University, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi An Jiao Tong University, Xi’an, Shanxi
  - Yuncheng Central hospital, Yuncheng, Shanxi
  - Chengdu Fifth Peoples Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Sichuan
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Shanghai East Hospital, Shanghai
- Czechia (30):
  - Medicus Services sro, Brandýs nad Labem
  - MUDr Libor Nechvatal sro, Brno
  - MUDr Karel Kamenik sro, Brno
  - Fakultni nemocnice Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - Edumed sro, Broumov
  - CorMedico sro, Bruntál
  - Dika centrum sro, Havirov - Mesto
  - Kardio Holesov sro, Holešov
  - Edumed sro, Hradec Králové
  - Edumed sro, Jaroměř
  - Kardiologie - Liberec sro, Liberec
  - Edumed sro, Náchod
  - PreventaMed sro, Olomouc
  - CCR Ostrava sro, Ostrava
  - MUDr Miroslav Koliba sro, Ostrava
  - Pratia Pardubice as, Pardubice
  - Kardiologie a Angiologie Praha sro - Komplexni Centrum Vyzkumu, Prevence a Lecby Kardiov Nemoci, Prague
  - Avicena - kardiologie, interna sro, Prague
  - Kardiologie Vinohrady sro, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Kardiologicke centrum MUDr Janky Skrobakove sro, Praha 5 - Smichov
  - MUDr Jarmila Otrubova, Prostějov
  - Kardio Vaclavik sro, Přerov
  - Nemocnice Slany, Slaný
  - Kardiologicka ambulance MUDr Ferkl, sro, Trutnov
  - Ansaldo sro, Uherské Hradiště
  - Clinical Trials Service sro, Uherské Hradiště
  - Kardiologicka Ambulance MUDr Michaela Cervinkova, sro, Ústí nad Labem
  - Kardiologie - Usti nad Labem sro, Ústí nad Labem
- Denmark (7):
  - Aarhus Universitetshospital, Aarhus N
  - Esbjerg sygehus Syddansk universitetshospital, Esbjerg
  - Frederiksberg/Bispebjerg Hospitaler, Frederiksberg
  - Herlev and Gentofte Hospital, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Hvidovre Hospital, Hvidovre
  - Sjaellands Universitetshospital, Roskilde, Roskilde
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Terveystalo Ruoholahti, Helsinki
  - Terveystalo Jyvaskyla, Jyväskylä
  - Turku University Hospital Tyks, Turku
- France (16):
  - Centre Hospitalier Universitaire Amiens Picardie - Site Sud, Amiens
  - Centre Hospitalier de Beziers, Béziers
  - Hospices Civils de Lyon Groupement Hospitalier Est - Hopital Louis Pradel, Bron
  - Centre Hospitalier Universitaire de Dijon - Hopital Francois Mitterrand, Dijon
  - Hopital prive Le Bois, Lille
  - Centre Hospitalier Régional Universitaire de Lille - Institut Coeur Poumon, Lille
  - Centre Hospitalier Universitaire de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital prive du Confluent, Nantes
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Saint Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier Intercommunal Toulon-La Seyne-sur-Mer - Hopital Sainte Musse, Toulon
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Centre Hospitalier de Tourcoing - Hopital Guy Chatiliez, Tourcoing
  - Centre Hospitalier Regional Universitaire de Tours - Hopital Trousseau, Tours
- Germany (28):
  - Rhoehn Klinik Campus Bad Neustadt, Bad Neustadt an der Saale
  - Segeberger Kliniken GmbH, Bad Segeberg
  - policum Berlin Friedenau, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Lippe, Detmold
  - Zentrum fuer klinische Pruefungen in der Facharztzentrum Dresden-Neustadt Betriebsgesellschaft, Dresden
  - Universitaetsklinikum Dresden, Dresden
  - ClinPhenomics CVC GmbH, Frankfurt am Main
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Medizinisches Versorgungszentrum im Altstadt-Carree Fulda, Fulda
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Cardiologicum Hamburg GbR, Hamburg
  - Kardiologische Praxis, Haßloch
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaetsklinikum Jena, Jena
  - Kardiopraxis Schirmer, Kaiserslautern
  - Universitaetsklinikum Leipzig, Leipzig
  - zero Praxen GbR, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - FutureMeds Offenbach, Offenbach
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Universitaetsklinikum Regensburg, Regensburg
  - Herz- und Gefaesszentrum Praxis Dr Overhoff Dr Kraemer, Siegen
  - Cardiologicum Herzklinik Ulm, Ulm
  - Praxis Dr med Ayham Al-Zoebi Facharzt fuer Innere Medizin und Kardiologie, Wermsdorf
- Greece (14):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Athens Naval Hospital, Athens
  - General Hospital for Thoracic Diseases of Athens "Sotiria, Athens
  - General Hospital of Athens Georgios Gennimatas, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - Alexandra Hospital, Athens
  - Attikon Hospital, Athens
  - General Hospital Asklipieio Voulas, Athens
  - General Hospital of Chios "Skilitsion", Chios
  - University Hospital of Larissa, Larissa
  - Hygeia Hospital, Marousi
  - General Hospital Of Nea Ionia Konstantopouleio Patision, Nea Ionia
  - Tzaneio General Hospital, Piraeus
  - Ahepa University Hospital, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Hungary (22):
  - Budapesti Szent Ferenc Korhaz, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Semmelweis Egyetem Varosmajori Sziv- es Ergyogyaszati Klinika, Budapest
  - Eszak-Pesti Centrum Korhaz - Honvedkorhaz, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Zugloi Egeszsegugyi Szolgalat, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Komaromi Selye Janos Korhaz, Komárom
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
  - Oroshazi Dr Laszlo Elek Korhaz es Rendelointezet, Orosháza
  - COROMED-SMO Kft, Pécs
  - DaVinci Maganklinika, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
  - Szegedi Tudomanyegyetem SZGYA Klinikai Kozpont Dr Bugyi Istvan Szentesi Multidiszciplinaris Centrum, Szentes
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Italy (13):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni xxiii, Bergamo
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia
  - Azienda Unita Sanitaria Locale Toscana sud est Ospedale S. Margherita, Cortona AR
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Azienda Unita Sanitaria Locale Romagna, Forlì
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliera di Rilievo Nazionale Specialistica dei Colli Monaldi, Napoli
  - Azienda Unita Sanitaria Locale Romagna, Rimini
  - ASL TO3 Ospedale di Rivoli, Rivoli
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
- Japan (19):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Sapporo, Hokkaido
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Tenyoukai Central Clinic, Kagoshima, Kagoshima-ken
  - Sagamihara Kyodo Hospital, Sagamihara-shi, Kanagawa
  - Kumamoto Kinoh Hospital, Kumamoto, Kumamoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - North Alps Medical Center Azumi Hospital, Kitaazumi-gun, Nagano
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Oita Red Cross Hospital, Ōita, Oita Prefecture
  - Fujinomiya City General Hospital, Fujinomiya-shi, Shizuoka
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu, Shizuoka
  - Medical Corporation Kenshinkai Minamino Cardiovascular Hospital, Hachioji-shi, Tokyo
  - Affiliated Central Clinic of Higashiyamato Hospital, Higashiyamato-shi, Tokyo
  - Tokyo Shinagawa Hospital Social Medical Corporation Association Tokyokyojuno-kai, Shinagawa-ku, Tokyo
  - NewHeart Watanabe Institute, Suginami-ku, Tokyo
  - Sanin Rosai Hospital, Yonago-shi, Tottori
- Netherlands (16):
  - Amsterdam Universitair Medisch Centrum, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Treant Zorggroep, locatie Scheper ziekenhuis Emmen, Emmen
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Frisius Medisch Centrum, locatie Leeuwarden, Leeuwarden
  - Ikazia Ziekenhuis, Rotterdam
  - D and A Research and Genetics, Sneek
  - Haga Ziekenhuis, The Hague
  - Zaans Medisch Centrum, Zaandam
- Poland (25):
  - Marek Dariusz Klimkiewicz Klimed Marek Klimkiewicz, Bialystok
  - Centrum medyczne intercore sp zoo, Bydgoszcz
  - American Heart of Poland Spolka Akcyjna, Chrzanów
  - Centrum Badan Klinicznych Agnieszka Mital, Elblag
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pawel Miekus, NZOZ Sopockie Centrum Badan Kardiologicznych ProCordis Pawel Miekus, Gdynia
  - Niepubliczny Zaklad Opieki Zdrowotnej Medica Jerzy Cygler, Giżycko
  - Pro Familia Altera Sp zoo, Katowice
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 2 Uniwersytetu Medycznego w Lodzi, Lodz
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Lodz
  - CenterMed Spzoo Centermed Lublin, Lublin
  - Szpital Swietej Anny w Miechowie, Miechów
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Olsztyn
  - Medicome Spolka z Ograniczona Odpowiedzialnoscia, Oświęcim
  - Centrum Medyczne Medyk Spolka z Ograniczona Odpowiedzialnoscia Spolka Komandytowa, Rzeszów
  - Velocity Skierniewice Spolka z Ograniczona Odpowiedzialnoscia, Skierniewice
  - Praktyka Lekarska Lidia Pawlowicz, Torun
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Tychy
  - Oha-Med Sp zoo, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Gabinet Lekarski Maciej Karcz, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Halina Serafin NZOZ Centrum Medyczne "Serafin-Med", Żarów
- Portugal (7):
  - Unidade Local de Saude de Almada-Seixal, EPE - Hospital Garcia de Orta, Almada
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Unidade Local de Saude do Alto Ave, EPE, Guimarães
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital Sao Francisco Xavier, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Unidade Local de Saude de Sao Joao, EPE - Hospital de Sao Joao, Porto
- Romania (10):
  - Cardioplus Center SRL, Baia Mare
  - cmi Cardiologie - Dr Pop Calin, Baia Mare
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed, Brasov
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Matcord Biomedica Buzau, Buzău
  - Consultmed SRL, Iași
  - Sal Med SRL, Piteşti
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - Cabinet Medical Individual Dr Podoleanu Cristian, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Slovakia (18):
  - Alian, sro, Bardejov
  - Narodny ustav srdcovych a cievnych chorob, as, Bratislava
  - Novate sro, Bratislava
  - Kardiomedina sro, Dolný Kubín
  - Nemocnica Dr Vojtecha Alexandra v Kezmarku no, Kežmarok
  - Medical group Kosice sro, Košice
  - Cardio D and R, sro Kosice, Košice
  - KardioLEV sro, Levoča
  - Kardio 1 sro, Lučenec
  - Nemocnicna as, Malacky
  - Oralek, sro, Námestovo
  - Kardiomed NZ, sro, Nové Zámky
  - KaCH, sro, Nové Zámky
  - Nemocnica Poprad, as, Poprad
  - Intermedis sro, Prešov
  - Medispol, sro, Prešov
  - Interna SK, sro, Svidník
  - Pentes, sro, Žilina
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (18):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario Arnau de Vilanova Lleida, Lleida, Catalonia
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Marina Salud de Denia, Denia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Sweden (8):
  - Falu Lasarett, Falun
  - Carlanderska sjukhuset, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Clemenstorgets Hjartmottagning, Lund
  - Vrinnevisjukhuset i Norrkoeping, Norrköping
  - Karolinska Universitetssjukhuset Solna, Solna
  - Capio Saint Gorans Hospital, Stockholm
  - Danderyds Sjukhus, Stockholm
- Switzerland (5):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Istituto Cardiocentro Ticino, Lugano
  - Kantonsspital Sankt Gallen, Sankt Gallen
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- Turkey (Türkiye) (7):
  - Afyonkarahisar Saglik Bilimleri Universitesi Hastanesi, Afyonkarahisar
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Mehmet Akif Ersoy Gogus Kalp ve Damar Cerrahisi Egitim ve Arastirma Hastanesi, Istanbul
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Necmettin Erbakan Universitesi Tip Fakultesi Hastanesi, Konya
- United Kingdom (12):
  - University Hospital Monklands, Airdrie
  - North Tyneside General Hospital, Ashington
  - Southmead Hospital, Bristol
  - St Richards Hospital, Chichester
  - Ninewells Hospital and Medicine School, Dundee
  - Royal Devon and Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Wycombe Hospital, High Wycombe
  - Highlands Clinical Research Facility, Raigmore Hospital, Inverness
  - University Hospital Crosshouse, Kilmarnock
  - University College London Hospital, London
  - Newcastle NIHR Commercial Research Delivery Centre, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this trial will be considered beginning 18 months after the trial has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this trial.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen trial/trials in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com